CLINICAL TRIAL: NCT00711594
Title: Phase I/II Open Label Trial of Continuous Once Daily Oral Treatment With BIBW 2992 - Phase I Trial in Advanced Non Small Cell Lung Cancer Patients & Phase II Trial in Non Small Cell Lung Cancer Patients Failing Erlotinib or Gefitinib.
Brief Title: LUX-Lung 4: BIBW 2992 (Afatinib) Phase I Trial in Advanced Non Small Cell Lung Cancer Patients & Phase II Trial in Non Small Cell Lung Cancer Patients Failing Erlotinib or Gefitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.33
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Results first posted 2013-11-13 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (2):
- BIBW 2992 MA2 (Experimental): Phase I step: Find maximum tolerated dose of the non-marketed substance:BIBW 2992 given orally. Escalating doses of BIBW 2992 starting at 20mg daily.
  Interventions: Drug: BIBW 2992 MA2 40mg/day; Drug: BIBW 2992 MA2 50mg/day; Drug: BIBW 2992 MA2 20mg/day
- BIBW 2992 QD (Experimental): Phase II step: Patients start continuous once daily oral treatment of BIBW 2992 at high dose, until progression or undue Adverse Events (AEs) develop. Patients can be dose-reduced up to two times if needed after temporary discontinuation of treatment due to drug-related AEs.
  Interventions: Drug: BIBW 2992 QD

INTERVENTIONS:
Drug: BIBW 2992 MA2 40mg/day — Phase I step: Increased dose cohorts from low dose to MTD
  Arms: BIBW 2992 MA2
Drug: BIBW 2992 MA2 50mg/day — Phase I step: Increased dose cohorts from low dose to MTD
  Arms: BIBW 2992 MA2
Drug: BIBW 2992 MA2 20mg/day — Phase I step: Increased dose cohorts from low dose to MTD
  Arms: BIBW 2992 MA2
Drug: BIBW 2992 QD — Phase II step: This is an open label study. Patients are treated with BIBW 2992 until disease progression or undue AEs.
  Arms: BIBW 2992 QD

SUMMARY:
The objective of the Phase I step is to estimate the MTD at a dose level up to 50 mg/day (i.e., overseas recommended Phase II dose) in patients with advanced NSCLC and to determine the recommended dose for the Phase II step.

The objective of the Phase II step is to estimate the efficacy of BIBW 2992 monotherapy in patients with first generation EGFR-TKI-resistant advanced NSCLC at the recommended dose determined in the Phase I step.

ELIGIBILITY:
Inclusion criteria:

Phase II step;

1. Patients with pathologic confirmation of NSCLC with tissue diagnosis or cytologic diagnosis, whose NSCLCs are locally advanced or metastatic Stage III-B / IV adenocarcinoma, and are inoperable and incurable with radiotherapy.
2. Patients who have received the following pretreatments for the treatment of relapsed or metastatic NSCLC.

   * Patients who have received at least one but not more than two lines of chemotherapy. ("Chemotherapy" means only the first line (doublet chemotherapies including a platinum) and/or the second line (single chemotherapy except for a platinum) of cytotoxic chemotherapy according to the standard chemotherapies, and erlotinib (Tarceva®) and gefitinib (Iressa®) should be excluded. One of the chemotherapy regimens must have been platinum-based. In addition, only one prior cytotoxic chemotherapy treatment regimen is allowed after adjuvant chemotherapy containing a platinum. More than two prior cytotoxic chemotherapy treatment regimens are not allowed.)
   * After the above chemotherapies, patients who once got clinical benefits (i.e. complete response, partial response or stable disease) but progressed following at least 12 weeks of treatment with erlotinib (Tarceva®) or gefitinib (Iressa®) as the most recent treatment. ("Clinical benefit" and "progression" should be confirmed by computed tomography (CT) or magnetic resonance imaging (MRI). In addition, "at least 12 weeks of treatment" should be 9 weeks or more as the actual "treatment period except for treatment pause due to adverse events and other reasons.) As long as the treatment is erlotinib or gefitinib monotherapy, patients can receive multiple regimens of either or both treatments, but one of the regimens should be for at least 12 weeks
3. Male or female patients age >=20 years at the enrolment.
4. Life expectancy of at least three (3) months after the start of administration of the investigational drug.
5. Eastern Cooperative Oncology Group (ECOG) performance Score 0 or 1.
6. Patients with at least one tumor lesion that can accurately be measured by CT or MRI in at least one dimension with longest diameter to be recorded as no less than double the slice thickness and >=10 mm.
7. Written informed consent that is consistent with ICH-GCP guidelines.

Exclusion criteria:

Phase II step;

1. Use of erlotinib (Tarceva®) or gefitinib (Iressa®) within two weeks before starting the study medication.
2. Patients who have received definitive thoracic radiotherapy with curative intent. Patients who have received radiotherapy or other investigational drugs (non-oncological) within four weeks before enrolment.
3. Significant gastrointestinal disorders with diarrhea as a major symptom e.g., Crohn's disease, mal-absorption, or CTCAE Grade >2 diarrhea of any etiology at the enrolment.
4. Patients with distinct / suspected pulmonary fibrosis or interstitial lung disease by the chest radiographic findings, or patients with a previous history of.
5. Brain tumor, and / or brain metastases, which are symptomatic or requiring treatment at the enrolment.
6. Other malignancies diagnosed within the past five years (other than carcinoma in situ of gastric cancer, colon cancer and cervical cancer, and non melanomatous skin cancer).
7. History of uncontrolled cardiac disease such as angina or myocardial infarction within the past 6 months at the enrolment, congestive heart failure including New York Heart Association (NYHA) functional classification of 3, or arrhythmia requiring treatment.
8. Coelomic fluid retention (such as pleural effusion, ascites or pericardial effusion) requiring treatment.
9. Uncontrolled concomitant diseases (e.g. diabetes mellitus, hypertension etc).
10. History of serious drug hypersensitivity.
11. Patients who do not have sufficient baseline organ function and whose laboratory data do not meet the following criteria at the enrolment.11

    * Haemoglobin count >=9.0 g/dL
    * Absolute neutrophil count (ANC) >=1500 / mm3
    * Platelet count >=100 000 / mm3
    * Serum creatinine <=1.5 mg/dL
    * Total bilirubin <=1.5 mg/dL
    * Aspartate aminotransferase (AST) and / or alanine aminotransferase (ALT) <=2.5x upper limit of normal range (if related to liver metastases <=2.5x upper limit of normal also)
    * PaO2 >=60torr or SpO2 >=92%
    * LVEF as measured by echocardiography or multigated blood pool imaging of the heart (MUGA scan) >=50%
    * QTc interval <0.47 second
12. Patients who disagree with using a medically acceptable method of contraception during the administration of the investigational drug and for at least 6 months after the end of administration.
13. Pregnant or breast-feeding women, or women suspected of being pregnant.
14. Known positive HBs antigen, HCV antibody, or HIV antibody test.
15. Known or suspected active drug or alcohol abuse.
16. Other patients judged ineligible for enrolment in the study by the investigator (sub-investigator).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (20):
- Japan (20):
  - 1200.33.010 Boehringer Ingelheim Investigational Site, Akashi, Hyogo
  - 1200.33.001 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1200.33.007 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1200.33.013 Boehringer Ingelheim Investigational Site, Hidaka, Saitama
  - 1200.33.011 Boehringer Ingelheim Investigational Site, Kanazawa, Ishikawa
  - 1200.33.003 Boehringer Ingelheim Investigational Site, Kashiwa, Chiba
  - 1200.33.019 Boehringer Ingelheim Investigational Site, Kobe, Hyogo
  - 1200.33.008 Boehringer Ingelheim Investigational Site, Koto-ku, Tokyo
  - 1200.33.020 Boehringer Ingelheim Investigational Site, Matsuyama, Ehime
  - 1200.33.006 Boehringer Ingelheim Investigational Site, Miyakojima-ku, Osaka
  - 1200.33.004 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1200.33.017 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1200.33.016 Boehringer Ingelheim Investigational Site, Niigata, Niigata
  - 1200.33.009 Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - 1200.33.005 Boehringer Ingelheim Investigational Site, Osaka-Sayama, Osaka
  - 1200.33.018 Boehringer Ingelheim Investigational Site, Sakai, Osaka
  - 1200.33.015 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1200.33.012 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1200.33.002 Boehringer Ingelheim Investigational Site, Sunto-gun, Shizuoka
  - 1200.33.014 Boehringer Ingelheim Investigational Site, Yufu, Oita

REFERENCES:
- [Derived] Katakami N, Atagi S, Goto K, Hida T, Horai T, Inoue A, Ichinose Y, Koboyashi K, Takeda K, Kiura K, Nishio K, Seki Y, Ebisawa R, Shahidi M, Yamamoto N. LUX-Lung 4: a phase II trial of afatinib in patients with advanced non-small-cell lung cancer who progressed during prior treatment with erlotinib, gefitinib, or both. J Clin Oncol. 2013 Sep 20;31(27):3335-41. doi: 10.1200/JCO.2012.45.0981. Epub 2013 Jul 1. PMID 23816963
- [Derived] Murakami H, Tamura T, Takahashi T, Nokihara H, Naito T, Nakamura Y, Nishio K, Seki Y, Sarashina A, Shahidi M, Yamamoto N. Phase I study of continuous afatinib (BIBW 2992) in patients with advanced non-small cell lung cancer after prior chemotherapy/erlotinib/gefitinib (LUX-Lung 4). Cancer Chemother Pharmacol. 2012 Apr;69(4):891-9. doi: 10.1007/s00280-011-1738-1. Epub 2011 Nov 10. PMID 22071596

RESULTS

PARTICIPANT FLOW:
Groups:
- BIBW 20mg: Continuous once daily oral treatment with BIBW 2992 20mg tablets
- BIBW 40mg: Continuous once daily oral treatment with BIBW 2992 40mg tablets
- BIBW 50mg (Phase I); BIBW 50mg (Phase II): Continuous once daily oral treatment with BIBW 2992 50mg tablets
Period: Overall Study
Arm/Group | BIBW 20mg | BIBW 40mg | BIBW 50mg (Phase I) | BIBW 50mg (Phase II)
Started | 3 | 3 | 6 | 62
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 6 | 62
Not completed — Progressive disease | 2 | 2 | 6 | 44
Not completed — Other Adverse Event | 1 | 0 | 0 | 16
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Until the snapshot for CTR
Groups:
- Total: Total of all reporting groups
Arm/Group | BIBW 20mg | BIBW 40mg | BIBW 50mg (Phase I) | BIBW 50mg (Phase II) | Total
Number analyzed (Participants) | 3 | 3 | 6 | 62 | 74
Age, Continuous [Median (Full Range); unit: years] — BIBW 20mg, 40mg, 50mg (Phase I)
  years | 65.0 [64 to 67] | 56.0 [46 to 57] | 63.0 [39 to 67] | 65.0 [33 to 84] | 65.0 [33 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 48 | 55
  Male | 1 | 1 | 3 | 14 | 19

OUTCOME MEASURES:

1. Primary Outcome: Phase I Step: Safety of BIBW 2992 Assessed Based on Incidence of Dose Limiting Toxicity (DLT) and Incidence & Intensity of Adverse Events According to CTCAE
Time Frame: start of treatment to end of treatment
Population: The "treated set" of patients was defined as all patients who received at least 1 dose of BIBW 2992 medication.
Measure: Number; unit: participants
Arm/Group | BIBW 20mg | BIBW 40mg | BIBW 50mg (Phase I)
Number analyzed (Participants) | 3 | 3 | 6
participants
  Patients with any AE | 3 | 3 | 6
  Investigator defined drug-related AEs | 3 | 3 | 6
  Other significant AEs (according to ICH E3) | 0 | 1 | 1
  AEs leading to discontinuation of trial drug | 1 | 0 | 0
  Serious AEs | 1 | 0 | 2
  SAE: Requiring hospitalisation | 0 | 0 | 1
  SAE: Prolonging hospitalisation | 1 | 0 | 1
  SAE: Other | 1 | 0 | 0
  Highest CTCAE grade for AEs (Grade 1) | 0 | 0 | 1
  Highest CTCAE grade for AEs (Grade 2) | 1 | 3 | 2
  Highest CTCAE grade for AEs (Grade 3) | 2 | 0 | 3
  Highest CTCAE grade for AEs (Grade 4) | 0 | 0 | 0
  Highest CTCAE grade for AEs (Grade 5) | 0 | 0 | 0
  Patients with any DLT (Course 1) | 0 | 0 | 1
  Patients with any DLT (All Courses) | 0 | 0 | 3

2. Primary Outcome: Phase II Step: Objective Tumour Response According to Response Evaluation Criteria in Solid Tumours (RECIST)
Description: The objective response (complete response [CR] and partial response [PR]) was defined as determined by the RECIST according to the best response to study treatment.
Time Frame: Tumour Assessment were performed at screening 14 days (prior to enrollment), in week 4, week 8, week 12 and in 8-week intervals thereafter, and at the end of trial visit (patients discontinuation), up to 41.3 months
Population: The "full analysis set" of patients was defined as all patients included in the treated set who have both baseline tumour imaging data and at least one analysable tumour imaging data after BIBW 2992 started.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIBW 50mg (Phase II)
Number analyzed (Participants) | 61
percentage of participants
  Independent review | 8.2 [2.7 to 18.1]
  Investigator assessment | 13.1 [5.8 to 24.2]

3. Secondary Outcome: Phase I Step: AUC0-24, AUCtau,ss of BIBW 2992 After Multiple Oral Administration
Description: area under the concentration-time curve of BIBW 2992 over the time interval 0-24 hours (AUC0-24), Area under the concentration-time curve of Afatinib in plasma at steady state (AUCtau,ss) after multiple oral administration Pharmacokinetic was abbreviated to PK.
Time Frame: AUC0-24: just before drug administration, 0:30,1:00, 2:00, 3:00, 4:00, 5:00, 7:00, 9:00, 24:00 on Day 1-2 in Course 1; AUCtau,ss: just before drug administration, 0:30,1:00, 2:00, 3:00, 4:00, 5:00, 7:00, 9:00, 24:00, 48:00, 72:00 on Day 28-31 in Course 1
Population: "Treated set" was defined as all patients who received at least 1 dose of BIBW2992. Some samples were excluded from calculation of descriptive statistics of plasma concentration because these were taken outside the allowed time-windows but used for calculation of PK parameters.
  Number of analyzed patients of BIBW 50mg:5(AUCtau,ss), 40mg:2(AUC0-24)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | BIBW 20mg | BIBW 40mg | BIBW 50mg (Phase I)
Number analyzed (Participants) | 3 | 3 | 6
ng·h/mL
  AUC0-24 | 147 (84.5) | 299 (6.01) | 539 (59.0)
  AUCtau,ss | 409 (16.5) | 1240 (9.73) | 1010 (71.5)

4. Secondary Outcome: Phase II Step: Clinical Benefit
Description: Clinical benefit was defined as a RECIST assessment of complete response, partial response, or stable disease according to the best response to study treatment as defined in the previous section. Clinical benefit presented as the disease control.
Time Frame: Tumour Assessment were performed at screening 14 days (prior to enrollment), in week 4, week 8, week 12 and in 8-week intervals thereafter, and at the end of trial visit (patients discontinuation) up to 41.3 months
Population: The "full analysis set" of patients was defined as all patients includes in the treated set who have both baseline tumour imaging data and at least one analysable tumour imaging data after BIBW 2992 started.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIBW 50mg (Phase II)
Number analyzed (Participants) | 61
percentage of participants
  Independent review | 65.6 [52.3 to 77.3]
  Investigator assessment | 72.1 [59.2 to 82.9]

5. Secondary Outcome: Phase II Step: Time to Objective Response
Description: Number of participants with first response at week 4, 8 and 12, assessed by investigator and independent review.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Number of patients
Arm/Group | BIBW 50mg (Phase II)
Number analyzed (Participants) | 61
Number of patients
  Time to first response (Week4, Independent) | 4
  Time to first response (Week8, Independent) | 1
  Time to first response (Week12, Independent) | 0
  Time to first response (Week4, Investigator) | 5
  Time to first response (Week8, Investigator) | 2
  Time to first response (Week12, Investigator) | 1

6. Secondary Outcome: Phase II Step: Duration of Objective Response
Description: Duration of objective response was defined as the time at which RECIST was first met for CR or PR (whichever was first recorded) until the first date that recurrent or progressive disease (PD) was objectively documented.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: weeks
Arm/Group | BIBW 50mg (Phase II)
Number analyzed (Participants) | 61
weeks
  Independent review | 19.9 [6.9 to 112.1]
  Investigator assessment | 16.1 [12.1 to 28.4]

7. Secondary Outcome: Phase I Step: Summary of Epidermal Growth Factor Receptor (EGFR) Mutation Findings
Time Frame: Screening visit
Population: The "treated set" of patients was defined as all patients who received at least 1 dose of BIBW 2992 medication.
Measure: Number; unit: participants
Arm/Group | BIBW 20mg | BIBW 40mg | BIBW 50mg (Phase I)
Number analyzed (Participants) | 2 | 3 | 6
participants
  Patients with positive EGFR mutation status | 2 | 1 | 2
  Del19 + T790M | 2 | 0 | 1
  L858R + T790M | 0 | 0 | 1
  S768I | 0 | 1 | 0

8. Secondary Outcome: Phase II Step: Duration of Clinical Benefit
Description: Presented as duration of disease control.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: Weeks
Arm/Group | BIBW 50mg (Phase II)
Number analyzed (Participants) | 61
Weeks
  Independent review | 19.9 [7.7 to 116.4]
  Investigator assessment | 20.9 [10.1 to 180.4]

9. Secondary Outcome: Phase II Step: Progression-free Survival (PFS)
Description: PFS was defined as the duration of time from the start of treatment until the day of objective tumour progression confirmed by tumour imaging (PD according to the RECIST) or death.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | BIBW 50mg (Phase II)
Number analyzed (Participants) | 61
Months
  Independent review | 4.5 [1.9 to 6.0]
  Investigator assessment | 4.6 [2.8 to 10.0]

10. Secondary Outcome: Phase II Step: Overall Survival (OS)
Description: OS was defined as the duration of time from the start of treatment to the time of death.
Time Frame: from start of treatment until end of follow up, up to 53 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | BIBW 50mg (Phase II)
Number analyzed (Participants) | 61
Months | 18.4 [11.9 to 36.3]

11. Secondary Outcome: Phase II Step: Safety of BIBW 2992 as Indicated by Intensity and Incidence of Adverse Events, Graded According to CTCAE
Description: outcome data show the number of patients with Adverse events (AE) by intensity and incidence of adverse events, graded according to CTCAE.
Time Frame: Start of treatment to end of treatment (up to 41.3 months) plus 4 week follow-up
Population: The "treated set" of patients was defined as all patients who received at least 1 dose of BIBW 2992 medication.
Measure: Number; unit: participants
Arm/Group | BIBW 50mg (Phase II)
Number analyzed (Participants) | 62
participants
  Patients with any AE | 62
  Investigator defined drug-related AEs | 62
  AEs leading to dose reduction of trial drug | 43
  AEs leading to discontinuation of trial drug | 19
  Serious AEs | 16
  SAE: Fatal | 1
  SAE: Immediate life-threatening | 1
  SAE: Requiring hospitalisation | 13
  SAE: Prolonging hospitalisation | 4
  SAE: Other | 1
  Highest CTCAE grade for AEs (Grade 1) | 0
  Highest CTCAE grade for AEs (Grade 2) | 11
  Highest CTCAE grade for AEs (Grade 3) | 48
  Highest CTCAE grade for AEs (Grade 4) | 2
  Highest CTCAE grade for AEs (Grade 5) | 1

12. Secondary Outcome: Phase II Step: Maximum CTC Grade During the Trial for Laboratory Parameters, Among Patients Who Experienced an Increase in CTC Grade From Baseline
Description: outcome data show the number of patients for the maximum CTC grade during the trial for laboratory parameters, among patients who experienced an increase in CTC Grade
Time Frame: Start of treatment to end of treatment (up to 41.3 months) plus 4 week follow-up
Population: The "treated set" of patients was defined as all patients who received at least 1 dose of BIBW 2992 medication.
  For activated partial thromboplastin time (APTT), N = 59 For Prothrombin Time and International Normalized Ratio (PT-INR), N = 61
Measure: Number; unit: participants
Arm/Group | BIBW 50mg (Phase II)
Number analyzed (Participants) | 62
participants
  White blood cell count (CTCAE Grade1) | 5
  White blood cell count (CTCAE Grade2) | 6
  White blood cell count (CTCAE Grade3) | 1
  White blood cell count (CTCAE Grade4) | 0
  White blood cell count (CTCAE Grade5) | 0
  Haemoglobin (CTCAE Grade1) | 21
  Haemoglobin (CTCAE Grade2) | 7
  Haemoglobin (CTCAE Grade3) | 1
  Haemoglobin (CTCAE Grade4) | 0
  Haemoglobin (CTCAE Grade5) | 0
  Platelets (CTCAE Grade1) | 4
  Platelets (CTCAE Grade2) | 0
  Platelets (CTCAE Grade3) | 0
  Platelets (CTCAE Grade4) | 0
  Platelets (CTCAE Grade5) | 0
  Neutrophils (CTCAE Grade1) | 20
  Neutrophils (CTCAE Grade2) | 5
  Neutrophils (CTCAE Grade3) | 1
  Neutrophils (CTCAE Grade4) | 0
  Neutrophils (CTCAE Grade5) | 0
  Lymphocytes (CTCAE Grade1) | 27
  Lymphocytes (CTCAE Grade2) | 7
  Lymphocytes (CTCAE Grade3) | 6
  Lymphocytes (CTCAE Grade4) | 0
  Lymphocytes (CTCAE Grade5) | 0
  APTT (CTCAE Grade1) | 1
  APTT (CTCAE Grade2) | 0
  APTT (CTCAE Grade3) | 0
  APTT (CTCAE Grade4) | 0
  APTT (CTCAE Grade5) | 0
  PT-INR (CTCAE Grade1) | 5
  PT-INR (CTCAE Grade2) | 0
  PT-INR (CTCAE Grade3) | 0
  PT-INR (CTCAE Grade4) | 0
  PT-INR (CTCAE Grade5) | 0
  Hypocalcaemia (CTCAE Grade1) | 16
  Hypocalcaemia (CTCAE Grade2) | 4
  Hypocalcaemia (CTCAE Grade3) | 0
  Hypocalcaemia (CTCAE Grade4) | 0
  Hypocalcaemia (CTCAE Grade5) | 0
  Hypernatraemia (CTCAE Grade1) | 1
  Hypernatraemia (CTCAE Grade2) | 0
  Hypernatraemia (CTCAE Grade3) | 0
  Hypernatraemia (CTCAE Grade4) | 0
  Hypernatraemia (CTCAE Grade5) | 0
  Hyponatraemia (CTCAE Grade1) | 14
  Hyponatraemia (CTCAE Grade2) | 0
  Hyponatraemia (CTCAE Grade3) | 1
  Hyponatraemia (CTCAE Grade4) | 0
  Hyponatraemia (CTCAE Grade5) | 0
  Hyperkalemia (CTCAE Grade1) | 8
  Hyperkalemia (CTCAE Grade2) | 2
  Hyperkalemia (CTCAE Grade3) | 1
  Hyperkalemia (CTCAE Grade4) | 0
  Hyperkalemia (CTCAE Grade5) | 0
  Hypokalemia (CTCAE Grade1) | 18
  Hypokalemia (CTCAE Grade2) | 0
  Hypokalemia (CTCAE Grade3) | 2
  Hypokalemia (CTCAE Grade4) | 0
  Hypokalemia (CTCAE Grade5) | 0
  AST/GOT, SGOT (CTCAE Grade1) | 12
  AST/GOT, SGOT (CTCAE Grade2) | 4
  AST/GOT, SGOT (CTCAE Grade3) | 0
  AST/GOT, SGOT (CTCAE Grade4) | 0
  AST/GOT, SGOT (CTCAE Grade5) | 0
  ALT/GPT, SGPT (CTCAE Grade1) | 8
  ALT/GPT, SGPT (CTCAE Grade2) | 7
  ALT/GPT, SGPT (CTCAE Grade3) | 1
  ALT/GPT, SGPT (CTCAE Grade4) | 0
  ALT/GPT, SGPT (CTCAE Grade5) | 0
  Alkaline phosphatase (CTCAE Grade1) | 14
  Alkaline phosphatase (CTCAE Grade2) | 1
  Alkaline phosphatase (CTCAE Grade3) | 0
  Alkaline phosphatase (CTCAE Grade4) | 0
  Alkaline phosphatase (CTCAE Grade5) | 0
  Creatine phosphatase (CTCAE Grade1) | 9
  Creatine phosphatase (CTCAE Grade2) | 4
  Creatine phosphatase (CTCAE Grade3) | 0
  Creatine phosphatase (CTCAE Grade4) | 0
  Creatine phosphatase (CTCAE Grade5) | 0
  Albumin (CTCAE Grade1) | 31
  Albumin (CTCAE Grade2) | 6
  Albumin (CTCAE Grade3) | 0
  Albumin (CTCAE Grade4) | 0
  Albumin (CTCAE Grade5) | 0
  Creatinine (CTCAE Grade1) | 13
  Creatinine (CTCAE Grade2) | 5
  Creatinine (CTCAE Grade3) | 2
  Creatinine (CTCAE Grade4) | 0
  Creatinine (CTCAE Grade5) | 0
  Uric acid (CTCAE Grade1) | 0
  Uric acid (CTCAE Grade2) | 0
  Uric acid (CTCAE Grade3) | 0
  Uric acid (CTCAE Grade4) | 2
  Uric acid (CTCAE Grade5) | 0
  Bilirubin, total (CTCAE Grade1) | 4
  Bilirubin, total (CTCAE Grade2) | 2
  Bilirubin, total (CTCAE Grade3) | 0
  Bilirubin, total (CTCAE Grade4) | 0
  Bilirubin, total (CTCAE Grade5) | 0
  Hyperglycaem (CTCAE Grade1) | 23
  Hyperglycaem (CTCAE Grade2) | 5
  Hyperglycaem (CTCAE Grade3) | 1
  Hyperglycaem (CTCAE Grade4) | 0
  Hyperglycaem (CTCAE Grade5) | 0
  Hypoglycaemia (CTCAE Grade1) | 2
  Hypoglycaemia (CTCAE Grade2) | 1
  Hypoglycaemia (CTCAE Grade3) | 0
  Hypoglycaemia (CTCAE Grade4) | 0
  Hypoglycaemia (CTCAE Grade5) | 0
  U. protein (qual) (CTCAE Grade1) | 20
  U. protein (qual) (CTCAE Grade2) | 6
  U. protein (qual) (CTCAE Grade3) | 0
  U. protein (qual) (CTCAE Grade4) | 0
  U. protein (qual) (CTCAE Grade5) | 0

13. Secondary Outcome: Phase II Step: Trough Plasma Concentrations of BIBW2992 After Multiple Oral Administration of BIBW 2992: Treatment course1 Day 15
Description: Outcome data show the geometric mean (gMean) of trough plasma concentrations of BIBW 2992 after multiple oral administration of BIBW.
  The dose determined from the result of the Phase I step (50 mg) will be used. Reduction of dose in accordance to the criteria specified by adverse events to 40 mg or 30 mg was possible.
Time Frame: Course 1 Day 15
Population: Plasma concentrations of BIBW2992 were to be presented for all patients and sampling points with concentrations above the lower limit of quantification. No patient was treated with 30 mg during the Course 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- BIBW 30mg: Continuous once daily oral treatment with BIBW 2992 30mg tablets
Arm/Group | BIBW 30mg | BIBW 40mg | BIBW 50mg (Phase II)
Number analyzed (Participants) | 0 | 5 | 49
ng/ml |  | 28.6 (33.2) | 44.0 (60.0)

14. Secondary Outcome: Phase II Step: Trough Plasma Concentrations of BIBW2992 After Multiple Oral Administration of BIBW 2992: Treatment course2 Day 1
Description: Outcome data show the gMean of trough plasma concentrations of BIBW 2992 after multiple oral administration of BIBW
Time Frame: Course 2 Day 1
Population: Plasma concentrations of BIBW2992 were to be presented for all patients and sampling points with concentrations above the lower limit of quantification.
  The dose determined from the result of the Phase I step (50 mg) will be used. Reduction of dose in accordance to the criteria specified by adverse events to 40 mg or 30 mg was possible.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | BIBW 30mg | BIBW 40mg | BIBW 50mg (Phase II)
Number analyzed (Participants) | 2 | 14 | 26
ng/ml | 27.2 (0.259) | 29.8 (47.8) | 38.3 (71.2)

15. Secondary Outcome: Phase II Step: Trough Plasma Concentrations of BIBW2992 After Multiple Oral Administration of BIBW 2992: Treatment course2 Day 15
Description: Outcome data show the gMean of trough plasma concentrations of BIBW 2992 after multiple oral administration of BIBW
Time Frame: Course 2 Day 15
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | BIBW 30mg | BIBW 40mg | BIBW 50mg (Phase II)
Number analyzed (Participants) | 5 | 18 | 16
ng/ml | 30.1 (24.8) | 32.1 (52.5) | 28.6 (138)

16. Secondary Outcome: Phase II Step: Summary of EGFR Mutation Findings
Time Frame: Screening visit
Population: The "treated set" of patients was defined as all patients who received at least 1 dose of BIBW 2992 medication.
Measure: Number; unit: participants
Arm/Group | BIBW 50mg (Phase II)
Number analyzed (Participants) | 62
participants
  EGFR Mutation test done (local or central) | 56
  Positive | 45
  Del19 | 22
  Del19 + L858R | 1
  Del19 + T790M | 1
  Del19 + Other | 1
  L858R | 15
  L858R + T790M | 1
  L858R + Other | 3
  L861Q | 1
  Negative | 11

17. Secondary Outcome: Phase I Step: Cmax,Cmax,ss of BIBW 2992 After Multiple Oral Administration
Time Frame: Just before start of the treatment to Course 4 Visit 4R2
Population: The "treated set" of patients was defined as all patients who received at least 1 dose of BIBW 2992 medication.Some samples were excluded from the evaluation because these were taken outside the allowed time-windows.
  Number of analyzed patients of BIBW 50mg cohort for Cmax,ss: 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BIBW 20mg | BIBW 40mg | BIBW 50mg (Phase I)
Number analyzed (Participants) | 3 | 3 | 6
ng/mL
  Cmax | 12.4 (101) | 18.9 (45.8) | 44.4 (60.6)
  Cmax,ss | 26.9 (24.9) | 83.3 (30.1) | 66.8 (71.6)

ADVERSE EVENTS:
Time Frame: from first administration of study medication up to 28 days after the completion of drug administration, up to 1260 days
Arm/Group | BIBW 20mg | BIBW 40mg | BIBW 50mg (Phase I) | BIBW 50mg (Phase II)
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/6 | 16/62
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIBW 20mg (N=3) | BIBW 40mg (N=3) | BIBW 50mg (Phase I) (N=6) | BIBW 50mg (Phase II) (N=62)
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIBW 20mg (N=3) | BIBW 40mg (N=3) | BIBW 50mg (Phase I) (N=6) | BIBW 50mg (Phase II) (N=62)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 1 | 10
Epidermolysis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 15
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 6 | 58
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1 | 0 | 9
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 24
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 3 | 40
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 17
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 18
Gait disturbance (General disorders) | 1 | 0 | 0 | 1
Malaise (General disorders) | 3 | 0 | 1 | 6
Mucosal dryness (General disorders) | 1 | 2 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 2 | 17
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 1 | 6
Tenderness (General disorders) | 1 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 6
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 7
Paronychia (Infections and infestations) | 1 | 2 | 3 | 42
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 2
Blood urine present (Investigations) | 0 | 0 | 3 | 5
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 2
Protein total decreased (Investigations) | 0 | 0 | 1 | 2
Weight decreased (Investigations) | 1 | 0 | 2 | 19
White blood cells urine positive (Investigations) | 2 | 0 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 3 | 37
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 11
Headache (Nervous system disorders) | 0 | 0 | 1 | 5
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 17
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 8
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 5 | 15
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 53
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 7
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 3
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.